CLINICAL TRIAL: NCT06324604
Title: Safety, Pharmacokinetics, and Pharmacodynamics of MTX-101 in Healthy Adults and Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mozart Therapeutics Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: MT-101-101
Record Dates: First submitted 2024-02-27; First posted 2024-03-22 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers; Celiac Disease; Type 1 Diabetes
Keywords: Healthy Volunteers; Celiac; Type 1 Diabetes
MeSH Terms: conditions — Celiac Disease; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Part A will enroll Healthy Adult Volunteers will be randomized, double-blind, placebo-controlled, single ascending dose (SAD), randomized to MTX-101 or placebo in a 1:1 ratio for the first 2 participants (sentinel dosing) and a 3:1 ratio thereafter. Participants in the multiple ascending dose (MAD) will be randomized in a 3:1 ratio and be dosed on Days 1 and 22.
  Part B of this study plans to enroll at least 24 (up to 44) participants with CeD or T1D, randomized in a 1:1 ratio, in 2 sequential cohorts. Approximately 12 CeD and 12 T1D patients will be enrolled in Part B, with the option to enroll up to a maximum of 44 total (CeD and/or T1D patients). Participants in Cohort B8 will be dosed with MTX-101 on Days 1 & 29, then placebo on Day 57 or placebo on Day 1 and MTX-101 on days 29 & 57. Participants in Cohort B9 will be dosed with MTX-101 or placebo on Day 1 and MTX-101 on Day 29. Patients will be followed for 6 months after the first dose.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort AS1 - Healthy Volunteers (Placebo Comparator): (n = 6): MTX-101, Dose level 1 IV or Placebo IV, Single dose
  Interventions: Drug: Placebo; Drug: MTX-101
- Cohort AS2 - Healthy Volunteers (Placebo Comparator): (n = 6): MTX-101, Dose Level 2 IV or Placebo IV, Single dose
  Interventions: Drug: Placebo; Drug: MTX-101
- Cohort AS3 - Healthy Vounteers (Placebo Comparator): (n = 6): MTX-101, Dose Level 3 IV or Placebo IV, single dose
  Interventions: Drug: Placebo; Drug: MTX-101
- Cohort AS4 - Healthy Volunteers (Placebo Comparator): (n =6): MTX-101, Dose Level 4 IV or Placebo IV, single dose
  Interventions: Drug: Placebo; Drug: MTX-101
- Cohort AS5 - Healthy Volunteers (Placebo Comparator): (n = 6): MTX-101, Dose level 6 IV or Placebo IV, Single Dose
  Interventions: Drug: Placebo; Drug: MTX-101
- Cohort AM1 - Healthy Volunteers (Placebo Comparator): Cohort AM1 (n = 6): MTX-101, Dose Level 5 IV or Placebo IV, dosed on Days 1 and 22 for a total of 2 doses
  Interventions: Drug: Placebo; Drug: MTX-101
- Cohort B8 - Celiac Disease or Type 1 Diabetes Patients (Placebo Comparator): * Dose Group 1 (n = 6): MTX-101 Dose Level 4 IV Day 1 and 29, placebo IV Day 57
  * Dose Group 2 (n = 6): Placebo IV Day 1, MTX-101 Dose Level 3 IV Day 29 and 57
  Interventions: Drug: Placebo; Drug: MTX-101
- Cohort B9 -Celiac Disease or Type 1 Diabetes Patients (Placebo Comparator): Dose Group 1 (n = 6): MTX-101 Dose Level 5 IV Days 1 and 29 Dose Group 2 (n = 6): Placebo IV Day 1, MTX-101 Dose Level 5 IV (or the maximum tolerated dose in Part A MAD) Day 29
  Interventions: Drug: Placebo; Drug: MTX-101

INTERVENTIONS:
Drug: Placebo — Placebo
Drug: MTX-101 — MTX-101 (bispecific CD8 Treg modulator)

SUMMARY:
First in human study to understand the potential side effects of MTX-101, how long MTX-101 lasts in the human body, and how MTX-101 affects specific human immune cells.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) study to evaluate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of MTX-101 in healthy adults (HA) and participants with celiac disease (CeD) and type 1 diabetes (T1D). This study will enroll HAs only in Part A and CeD and T1D patients only in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age ≥ 18 and ≤ 65 years at the time of anticipated dosing (Day 1).
* Healthy individuals without known current or chronic medical conditions, including no history of any autoimmune diseases, in the opinion of the Investigator.
* Body mass index (BMI) ≥ 18 kg/m2 and ≤ 32 kg/m2.
* Body weight ≥ 45and ≤ 100 kg.
* Negative Coronavirus Disease 2019 (COVID-19) test within 24 hours prior to each dose.
* Persons of child-bearing potential must have a negative pregnancy test and either abstain from sex or use highly effective method(s) of birth control from Day 1 through the duration of the study.

Exclusion Criteria:

* Clinically significant findings in physical examination (PE), vital signs (blood pressure, heart rate, and body temperature), electrocardiogram (ECG), and safety laboratory parameters at Screening in the opinion of the Investigator.
* Renal function calculated by the Chronic Kidney Disease-Epidemiology (CKD-EPI) equation with estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73 m2 or abnormal level of proteinuria detected by dipstick at the time of Screening.
* Any disease or condition that, in the opinion of the Investigator, might significantly compromise the cardiovascular, hematological, renal, hepatic, pulmonary (including chronic asthma), endocrine (e.g., diabetes), central nervous, or gastrointestinal (including an ulcer) systems.
* Receipt of an investigational drug within 28 days or 5 half-lives (whichever is longer) of the investigational drug(s) prior to Day 1.
* Positive serology for human immunodeficiency virus (HIV) type 1 or 2, hepatitis (Hep) B surface antigen, or Hep C.
* Positive test results for drug screen, including alcohol, at the time of Screening or on Day 1 prior to randomization.
* Use of tobacco or nicotine-containing products more than the equivalent of 5 cigarettes/week within 30 days prior to (first) dosing.

Participants must abstain from nicotine use while inpatient.

* History of receiving a live vaccine within 1 month of Screening.
* History of splenectomy.
* History of COVID or influenza vaccine within 2 weeks prior to Screening.
* Planning to receive any vaccinations during the study period.
* History of recurrent infections of uncertain cause.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Safety of single, ascending dose levels of MTX-101 | Enrollment to 8 weeks post dose
  Assess the safety of single, ascending dose levels of MTX-101 by evaluating the incidence, severity, and seriousness of treatment-emergent adverse events
Safety of multiple, ascending dose levels of MTX-101 | Enrollment to 11 weeks following the last dose
  Assess the safety of multiple, ascending dose levels of MTX-101by evaluating the incidence, severity, and seriousness of treatment-emergent adverse events

SECONDARY OUTCOMES:
pharmacokinetics (PK) of MTX-101 | Enrollment to 11 weeks following the last dose
  Characterize the pharmacokinetics (PK) of MTX-101 by measuring the maximum time of occurrence for maximum plasma drug concentration (Cmax)
pharmacokinetics (PK) of MTX-101 | Enrollment to 11 weeks following the last dose
  Characterize the pharmacokinetics (PK) of MTX-101 by measuring the time of occurrence for maximum plasma drug concentration (Tmax).
pharmacokinetics (PK) of MTX-101 | Enrollment to 11 weeks following the last dose
  Characterize the pharmacokinetics (PK) of MTX-101 by measuring the maximum plasma drug concentration (Cmax), minimum plasma drug concentration (Cmin), and area under the plasma drug concentration versus time curve from time 0 to last measurable concentration (AUC(0-t))
anti-drug antibody (ADA) formation | Enrollment to 11 weeks following the last dose
  Evaluate incidence of anti-drug antibody (ADA) formation by measuring the detect the presence of anti-MTX-101 antibodies in participant's blood.

OTHER OUTCOMES:
pharmacodynamics (PD) of MTX-101 | Enrollment up to 11 weeks following the last dose
  Evaluate how MTX-101 affect the immune system by the measuring the activity, presence and amount of signaling proteins and cells that help control inflammation.
Receptor occupancy of MTX-101 | Enrollment up to 11 weeks following the last dose
  To examine the binding ability of MTX-101 to targets on the cell surface.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (3):
  - Wesley Research Institute, Auchenflower, Queensland
  - Nucleus Network Brisbane, Herston, Queensland
  - The Royal Melbourne Hospital, Melbourne, Victoria
- Eastern Health; Box Hill Hospital, Box Hill, Victoria, Austria

IPD SHARING:
Plan to Share IPD: Undecided